CLINICAL TRIAL: NCT05839548
Title: Articaine Efficacy and Safety for 3 Years Old Children: a Clinical Randomized Control Trial
Brief Title: Articaine Efficacy and Safety for 3 Years Old Children
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qassim Health Cluster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 607\43\7809
Record Dates: First submitted 2023-03-16; First posted 2023-05-03 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Dental Caries in Children; Dental Diseases; Pulp Disease, Dental; Behavior, Child
Keywords: Articaine.; Local anaesthesia.; Child.; Pain.
MeSH Terms: conditions — Stomatognathic Diseases; Dental Pulp Diseases; Child Behavior; Pain | interventions — Mepivacaine; Epinephrine; Carticaine

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, clinical trial with two parallel arms, to evaluate the safety and efficacy of 4% Articaine, 2% Mepivacaine on vital and non-vital primary teeth that needs restorative, pulp therapy, or dental extraction by using buccal infiltration technique. The effect will be assessed by measuring the pain experience during injection and treatment procedures, and by assessing the child's behavior during the procedure, and postoperative pain and complications. The study consisted of a screening period for up to 6 months. A Qualified participants through the screening assessments will be assigned randomly to receive either 4% Articaine, or 2% Mepivacaine.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2% Mepivacaine with epinephrine 1:100,000. (Active Comparator): Brand Name: 2% Medicaine with epinephrine 1:100,000.
  Interventions: Drug: Mepivacaine 2% with epinephrine 1:100,000
- 4% Articaine with epinephrine 1:100,000 (Experimental): Brand Name: 4% Septanest with epinephrine 1:100,000.
  Interventions: Drug: Articaine (4%) with epinephrine 1:100,000

INTERVENTIONS:
Drug: Mepivacaine 2% with epinephrine 1:100,000 — Local Anesthesia
  Other Names: medicaine 2%
  Arms: 2% Mepivacaine with epinephrine 1:100,000.
Drug: Articaine (4%) with epinephrine 1:100,000 — Local Anesthesia
  Other Names: septanest 4%
  Arms: 4% Articaine with epinephrine 1:100,000

SUMMARY:
The primary purpose of this study is to determine the local anesthetic efficacy and safety of 4% Articaine compared 2% Mepivicaine in 3 years old children, by using infiltration technique for primary teeth that required restorative, pulp therapy, or dental extraction procedure, as assessed by measuring the pain experience during injection and treatment procedures, child's behavior during the procedure, and postoperative complications.

DETAILED DESCRIPTION:
Articaine has been widely used in dental surgery. Dentists started to use carticaine around 1977. In dentistry, articaine has been investigated extensively. Clinical trials comparing articaine mostly with lidocaine have varied in study design and site of action. The overwhelming majority of references in the literature describing the alleged neurotoxicity of articain concern paraesthesia and prolonged numbness after dental procedures. An excellent review of the dental literature was published last year. The authors concluded that articaine is a safe and effective local anesthetic drug to use in all aspects of clinical dentistry for patients of all ages, with properties comparable to other common local anesthetic agents. Although there may be controversy regarding its safety and advantages in comparison to other local anesthetics, there is no conclusive evidence demonstrating neurotoxicity or significantly superior anesthetic properties of articaine for dental procedures. The choice whether to use articaine or another local anesthetic is based on the personal preference and experiences of individual clinicians. 3Currently, articaine is available as a 4% solution containing 1:100,000 or 1:200,000 epinephrine. Clinical trials comparing 4% with 2% solutions show no clinical advantage of 4% over a 2% solution.

ELIGIBILITY:
Inclusion criteria:

All patients have to meet all of the following inclusion criteria. They are eligible if:

1. They are Healthy (ASA 1: no acute or chronic disease, normal BMI percentile for age.

1. They are 36 to 47 months old children.
2. Intellectually qualified for communication.
3. They have under gone either clinically indicated gingival abscess, dental caries or pathological root resorption or periapical radiolucency showing on the radiograph.
4. Child's body weight at least 15 kg.
5. Ability to communicate effectively in the Arabic or English language.
6. Not taking any agents likely to interfere with reporting of pain (analgesics).
7. Needs any of the following procedure: Class I cavity, Class II cavity, pulpotomy, pulpectomy, stainless steel crown (SSC) or extraction.
8. Prior to enrollment, all radiographic data must be found acceptable by pediatric dentist.
9. Written and singed informed consent from legally acceptable representative.

Exclusion criteria:

Patients are excluded from the study if:

1. Patients have allergic to local anesthetic with epinephrine (sulphites or amide).
2. Intellectual or severe emotional problems. patient with intellectual development is significantly lower than average and his or her ability to adapt to the environment is consequently limited like autism, Down syndrome, fragile x syndrome, fetal alcohol syndrome, and Prader-Willi syndrome.
3. Considerable behavior problems.
4. Parents refuse participation in the trial.
5. History of previous bad dental experience.
6. Primary tooth who had a history of failed pulp therapy.
7. They have uncontrolled medical condition.
8. They use immunosuppressive agents, rifampin, or anticonvulsants, or any other medication.
9. Glucose 6 phosphate dehydrogenase deficiency.
10. Congenital cardiac diseases.
11. Seizures or uncontrolled epilepsy.

Ages: 36 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure (mmHg). | 5 minutes before, during, and after 30 minutes of dental procedure.
  Normal blood pressure, defined as a systolic pressure less than 120, and a diastolic pressure less than 80.
Change in pulse rate (beats per minute). | 5 minutes before, during, and after 30 minutes of dental procedure.
  Pulse rate is the frequency of the heartbeat measured by the number of contractions of the heart per minute.
Change in respiratory rate (breaths per minute). | 5 minutes before, during, and after 30 minutes of dental procedure.
  The respiration rate is the number of breaths a person takes per minute.
Dental pain assessment: Frankl Behavior Rating Scale (FBRS). | up to 30 minutes after dental procedure.
  Frankl Behavior Rating Scale (FBRS) dichotomized into definitely negative (1), negative (2), positive (3), definitely positive (4).
Dental pain assessment: Faces, Legs, Activity, Cry, and Consolability. (FLACC). | up to 30 minutes after dental procedure.
  Each category is scored on the 0-2 scale, which results in a total score of 0-10. 0: relaxed and comfortable,1-3: mild discomfort, 4-6: moderate discomfort, 7-10: sever discomfort or pain or both.

SECONDARY OUTCOMES:
Post-operative complications. | 24 hours after dental procedure.
  asking the parent in next 24 hours from dental procedure, by using parents' post operative pain measure (PPPM). It will be dichotomized into absent (0-5) and present (6-15).

CONTACTS AND LOCATIONS:
Overall Officials: Murad A. Alrashdi, ABPD, Study Chair — Qassim University; Asya A. Almansour, SBPD, Principal Investigator — Ministry of Health, Qassim cluster.; Atyaf A. Alhunti, Study Director — Qassim University
Locations (1):
- Qassim University, Burayadh, Al-Qassim Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elheeny AAH. Articaine efficacy and safety in young children below the age of four years: An equivalent parallel randomized control trial. Int J Paediatr Dent. 2020 Sep;30(5):547-555. doi: 10.1111/ipd.12640. Epub 2020 Apr 13. PMID 32223002
- [Background] Brignardello-Petersen R. Articaine and lidocaine probably have similar effects in 3- to 4-year-old children undergoing pulpotomy of a primary molar. J Am Dent Assoc. 2020 Oct;151(10):e93. doi: 10.1016/j.adaj.2020.06.029. Epub 2020 Aug 11. No abstract available. PMID 32797942
- [Background] Massignan C, Silveira Santos P, Cardoso M, Bolan M. Efficacy and adverse events of 4% articaine compared with 2% lidocaine on primary molar extraction: A randomised controlled trial. J Oral Rehabil. 2020 Aug;47(8):1031-1040. doi: 10.1111/joor.12989. Epub 2020 May 25. PMID 32383196
- [Background] Rayati F, Haeri M, Norouziha A, Jabbarian R. Comparison of the efficacy of 4% articaine with epinephrine 1:100,000 and 2% lidocaine with epinephrine 1:100,000 buccal infiltration for single maxillary molar extraction: a double-blind, randomised, clinical trial. Br J Oral Maxillofac Surg. 2021 Jul;59(6):695-699. doi: 10.1016/j.bjoms.2020.09.009. Epub 2020 Sep 11. PMID 34053801
- [Derived] Alrashdi M, Alhunti A, Almansour A. Efficacy and safety of articaine in 3-year-old children for dental procedures: a protocol for a clinical randomised control trial in Saudi Arabia. BMJ Open. 2023 Oct 21;13(10):e077751. doi: 10.1136/bmjopen-2023-077751. PMID 37865418